CLINICAL TRIAL: NCT00666471
Title: Minimally Invasive Control of Epistaxis: Efficacy and Economic Analysis
Brief Title: Minimally Invasive Control of Epistaxis (MICE)
Acronym: MICE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: one PI (BM) no longer felt he had clinical equipoise regarding the intervention. No adverse events.
Sponsor: University of Calgary (Other)
Responsible Party: Joseph C. Dort MD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCENT0002
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Epistaxis
Keywords: epistaxis; Epistaxis refractory to emergency physician treatment
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MICE
  Interventions: Procedure: MICE
- 2 (Active Comparator): SPA ligation
  Interventions: Procedure: SPA ligation

INTERVENTIONS:
Procedure: MICE — MICE
  Arms: 1
Procedure: SPA ligation — SPA ligation
  Arms: 2

SUMMARY:
Epistaxis is a common disorder with 60% of the population suffering from one episode and 10% of these cases requiring medical attention. Between March 2006 and March 2007, in Calgary, Alberta, there were 1500 presentations of epistaxis to adult emergency rooms with 7% of these (105 patients) requiring packing with admission. Common methods to control epistaxis include, nasal packing (88%), operative arterial ligation (10%), and arterial embolization (2%). A cost analysis demonstrated that nasal packing had a lower cost compared to embolization and arterial ligation, and all modalities had similar lengths of stay (Goddard, Otolaryng Head Neck Surg. 2006). Arterial ligation is the current recommended therapy for recurrent or refractory epistaxis, with a success rate of 98%. With the advancement of endoscopic techniques, emergency room Minimally Invasive Control of Epistaxis (M.I.C.E.) allows for selective packing and cauterization, which provides the patient with retained function of their nasal cavity and prevents a hospital admission, resulting in significant cost savings.

Hypothesis:

Does the M.I.C.E. procedure provide significant cost savings compared to operative sphenopalatine artery ligation? Null hypothesis is that there is no difference in hospital admission rates between M.I.C.E. and operative sphenopalatine artery ligation.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old, Presenting to Rockyview General Hospital Emergency room
* No coagulopathy (must have INR reversed before inclusion)
* Available for follow-up at 1 week and 1 month in Calgary, Alberta
* Refractory or Recurrent Epistaxis defined as:

  * Refractory = unable to control epistaxis with bilateral Merocel™ Nasal Tampons fully inserted into nasal cavity
  * Recurrent = epistaxis after removal of Merocel™ Nasal Tampons following outpatient packing for 48 hours

Exclusion Criteria:

* Uncorrectable coagulopathy
* Unable to comply with procedure
* Pregnancy
* Non-Calgary emergency room presentation
* Severe posterior epistaxis requiring intubation for airway protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in hospital admission requirement between M.I.C.E. and Operative Sphenopalatine Ligation | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rockyview General Hospital / University of Calgary, Calgary, Alberta, Canada